CLINICAL TRIAL: NCT04157309
Title: Alternating Cycle / Direct Confirmation Redox Project (AC/DC)
Brief Title: Alternating Urine Redox Status Of Consecutive Menstrual Cycles
Acronym: ACDC
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Urobiologics LLC (Unknown)
Responsible Party: Principal Investigator, Daniel McConnell, Associate Research Scientist, University of Michigan
Other Study IDs: HUM00171526
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Pregnancy Related; Gender
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will involve the collection and analysis of urine samples from non-pregnant women to determine the existence of alternating redox status between two consecutive menstrual cycles.

DETAILED DESCRIPTION:
The Sponsor believes there is variability in the relative redox status in women's urine across menstrual cycles. This validation study will involve the collection and analysis of urine samples from non-pregnant women to determine the existence of alternating redox status between two consecutive menstrual cycles. If the hypothesis is proved, future research could examine if there are related fertility issues.

ELIGIBILITY:
Inclusion Criteria:

1. Female subject, between the years 18-30, at the time of consent.
2. Subject is willing to participate and is capable of giving informed consent. (Note: Consent must be obtained prior to any study-related procedures.)
3. Subject must be willing to comply with all study procedures and must be available to participate for the duration of the study.
4. Subject agrees to avoid alcohol, unapproved medications (prescription, OTC, or other), marijuana products, and illicit substances for 3 days prior to each urine collection.

Exclusion Criteria:

* 1. Subject is pregnant, or trying to or planning to become pregnant during the study.

  2. Subject was pregnant within 1 year of beginning study, regardless of the outcome of pregnancy.

  3. Subject who is breastfeeding. 4. Subject who is not menstruating for any reason or plans to undergo or change circumstances that might affect menstruation (e.g., certain athletic training regimens, significant dietary changes).

  5. History of recent or current irregular menstrual cycles (as self-reported by the subject).

  6. Subject reports she has been told by a medical professional that she is not ovulating (i.e., has anovulatory periods) at any time during the previous 12 months.

  7. Subject is using or planning to use any method to regulate her periods. 8. Subject smokes (includes tobacco and marijuana) or vapes. 9. By history, subject has medical problems that might influence the results of the study, such as endocrinologic, renal, or hormonal problems.

  10. Known polycystic ovarian syndrome (by history). 11. Subject is taking or planning to take hormones or hormone- enhancing/manipulating pharmaceuticals (including "morning after pill" [levonorgestrel], birth control pills, Clomid [clomiphene citrate], Femara [letrozole], Cialis [tadalafil]*, Viagra [sildenafil]* and similar medications) and/or agents to influence hormonal status such as herbal products or nutritional supplements. (*Not approved for use and should be avoided by women.) 12. Subject is using or planning to use hormonal contraceptives of any type, including oral contraceptives and intrauterine devices.

  13. Subject is using or planning to use hormonal therapies for acne vulgaris or other conditions, including spironolactone, flutamide, metformin, or oral contraceptives used as acne therapies, including Ortho Tri-Cyclen (combination of norgestimate and ethinyl estradiol [EE]), Estrostep (combination of norethindrone acetate and EE), and Yaz/Yasmin (combination of drospirenone and EE).

  14. Subject is using or planning to use estrogen products, including topicals/creams, for any purpose.

  15. Subject is using or planning to use androgens or anabolic steroids (e.g., stanazolol/danazol) for any reason, including for training or athletic purposes..

  16. Subject has attempted or taken IVF or IUI treatment within the prior six months.

  17. Subject has uncontrolled diabetes or other significant medical disorder that might, in the investigator's opinion, preclude completion of the study or suggest that an exclusion criterion will ensue.

  18. Subject reports difficulty handling biologic fluids, specifically urine, or gives other reasons why she is hesitant to participate.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — eligibility requires the subject to be a normally cycling female
Study Population: Approximately 40 women with normal reported menstrual cycles will be included in this validation study.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-01-04 (Actual); Study Completion 2021-01-04 (Actual)

PRIMARY OUTCOMES:
Redox potential of urine | 12 months
  The redox potential will be measured over two consecutive cycles to determine the variability in the relative redox status in women's urine.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Ellis, Study Director — University of Michigan; Kuldeep Veerma, Study Director — Urobiologics LLC
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT04157309/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT04157309/ICF_001.pdf